CLINICAL TRIAL: NCT07385287
Title: Randomized, Double-Blind, Placebo-Controlled Trial to Assess Safety, Immunogenicity, and Protective Efficacy Against Naturally Transmited Plasmodium Falciparum Malaria of One and Two Dose Regimens of a Late Liver Stage-arresting, Replication-competent Plasmodium Falciparum Sporozoite Vaccine (Sanaria® PfSPZ-LARC2 Vaccine) in Healthy Malaria-Exposed Adults in Burkina Faso
Brief Title: Phase 2 Field Trial of PfSPZ-LARC2 Vaccine in Burkinabe Adults
Acronym: BFSPZL2
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanaria Inc. (Industry)
Collaborators: University of Maryland, Baltimore (Other); Seattle Children's Hospital (Other); University of California, Los Angeles (Other); Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BFSPZL2; 6003.04 (Other Grant/Funding Number: Gates Foundation)
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Malaria (Plasmodium Falciparum)
Keywords: malaria; Plasmodium falciparum; PfSPZ Vaccine; PfSPZ-LARC2 Vaccine
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor's clinical and regulatory teams
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 2 SIngle Dose Vaccine Group (Experimental): Group 2: one dose of normal saline placebo and one dose of PfSPZ-LARC2 Vaccine (6x10^5 PfSPZ) four weeks apart.
  Interventions: Biological: Genetically attenuated PfSPZ Vaccine; Other: Normal Saline (0.9% Sodium Chloride)
- Group 1 Double Dose Vaccine Group (Experimental): Group 1: two doses of PfSPZ-LARC2 Vaccine (4x10^5 PfSPZ) four weeks apart.
  Interventions: Biological: Genetically attenuated PfSPZ Vaccine
- Group 3 Placebo (Placebo Comparator): Group 3: two doses of normal saline placebo four weeks apart.
  Interventions: Other: Normal Saline (0.9% Sodium Chloride)

INTERVENTIONS:
Biological: Genetically attenuated PfSPZ Vaccine — PfSPZ-LARC2 Vaccine is composed of aseptic, purified, vialed, cryopreserved, genetically altered PfNF54 sporozoites (SPZ). After thawing, the vaccine is diluted in phosphate buffered saline (PBS) with human serum albumin (HSA) to achieve the correct dosage and is administered by direct venous inoculation (DVI) into a superficial arm or hand vein within 30 minutes of thaw. PfSPZ-LARC2 Vaccine is manufactured by the trial sponsor, Sanaria Inc.
  Arms: Group 1 Double Dose Vaccine Group; Group 2 SIngle Dose Vaccine Group
Other: Normal Saline (0.9% Sodium Chloride) — The placebo control is normal saline solution (0.9% sodium chloride), purchased commercially from Pfizer, and is also administered by DVI.
  Arms: Group 2 SIngle Dose Vaccine Group; Group 3 Placebo

SUMMARY:
This is a Phase 2 clinical trial of Plasmodium falciparum (Pf) late liver stage-arresting replication-competent (LARC) sporozoite (SPZ) vaccine (Sanaria® PfSPZ-LARC2 Vaccine). It represents the next step in the development of this vaccine toward licensure, following a successful Phase 1 program in which the vaccine was shown to be safe (fully attenuated), well tolerated and immunogenic in malaria-exposed 1- to 45-year-olds in Burkina Faso (BFSPZL1 trial) and in malaria-naive adults in the US (USSPZL1 trial). Protection data will be available in March 2026 from the USSPZL1 trial, but these data will be from malaria-naive adults undergoing controlled human malaria infection (CHMI), representing (1) a different population with respect to immune status compared to malaria-exposed African adults, and (2) a one-time malaria exposure to a single malaria strain, compared to the ongoing, heterogeneous infection risk in nature. It is therefore important to assess field efficacy in Africa as soon as possible, to ascertain the potential value of PfSPZ-LARC2 Vaccine in addressing the World Health Organization's (WHO's) call for vaccines with high efficacy (>90%) against Pf infection naturally transmitted in endemic populations, with a focus on high burden sub-Saharan countries. PfSPZ-LARC2 Vaccine is especially promising because of data in malaria-naive adults showing that a biosimilar LARC vaccine called GA2 (aka LARC1) provided 90% vaccine efficacy (VE) against CHMI after administration of a single dose by mosquito bite, as recently published by the Leiden University Medical Center.

The PfSPZ comprising PfSPZ-LARC2 Vaccine contain a double deletion of the genes encoding the Mei2 and LINUP proteins, both of which are required for transition from liver to blood stage malaria. As a result, mei2-/linup- parasites undergo developmental arrest in the late liver stages without releasing merozoites into the blood stream. No blood stage parasites are produced, either asexual or sexual, and the parasite life cycle does not progress. Because Pf parasites with the LARC phenotype replicate in the liver before disintegrating, they amplify and diversify parasite protein expression and are expected to be a potent immunogen to induce anti-malarial immunity, equaling or exceeding the potency and efficacy of the replication-competent chemo-attenuated Sanaria® PfSPZ-CVac (chloroquine) vaccine approach. Because the parasites are intrinsically attenuated, they are expected to be safe and well tolerated, similar to radiation-attenuated Sanaria® PfSPZ Vaccine, to the replication deficient, early arresting PfSPZ-GA1 Vaccine, and to the single-gene(mei2)-deleted GA2 (LARC1) parasites tested at the Leiden University Medical Center that provided 90% protection against CHMI after a single dose as described above. In summary, the late liver stage arresting replication competent, genetically attenuated PfSPZ-LARC2 Vaccine should combine the best-in-class immunogenic potency and protective efficacy of replicating PfSPZ-CVac (chloroquine) with the excellent safety and tolerability of the early arresting, non-replicating radiation attenuated PfSPZ Vaccine, genetically attenuated PfSPZ-GA1 Vaccine, and genetically attenuated GA2 vaccine.

High level efficacy against naturally transmitted Pf in this trial will set the stage for Phase 3 testing and licensure. It will be complimentary to data from other planned trials to establish the following target populations: 1) women of child-bearing potential and pregnant women, to prevent pregnancy malaria; 2) children, to prevent pediatric malaria; and, eventually, 3) entire populations, to halt transmission and achieve regional malaria elimination. This development path aimed at endemic populations is being pursued in parallel with studies in malaria-naive individuals aiming to concurrently license a high efficacy malaria vaccine for travelers from non-malaria endemic to malaria-endemic areas.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, single-center Phase 2 clinical trial. Healthy nonpregnant, non-lactating adults will be enrolled. Women of child-bearing potential must agree to high efficacy birth control during the period of immunization. Screening tests will include an ECG, hepatitis B and C serology, HIV testing, sickle cell testing, a thick blood smear (TBS), white blood count, neutrophil count, lymphocyte count, hemoglobin, platelets, creatinine, alanine aminotransferase (ALT), bilirubin, gamma-glutamyl transferase (GGT) and a fasting blood glucose for all screenees to assure overall good health, and a pregnancy test for women.

The trial will compare a single dose regimen (6x10^5 PfSPZ administered once) to a two dose regimen (4x10^5 PfSPZ administered twice). There are three groups:

Group 1: two doses of PfSPZ-LARC2 Vaccine (4x10^5 PfSPZ) four weeks apart. Group 2: one dose of normal saline placebo and one dose of PfSPZ-LARC2 Vaccine (6x10^5 PfSPZ) four weeks apart.

Group 3: two doses of normal saline placebo four weeks apart. All participants will be cleared of any existing parasitemia by (minimally) a three day treatment course of artemether /lumefantrine. This will be done 5-6 weeks prior to the first dose of investigational product, to prevent the known immunosuppressive effects of parasitemia on the induction of protective immunity and to prevent such infections from recrudescing later in the trial. If, at a pre-immunization visit 2 weeks before the first dose, any participant is positive by TBS, they will be retreated with the same regimen of artemether/lumefantrine. Clearance will be repeated 2 weeks before the second dose in all participants. The justification for assuring TBS negative status prior to each immunization is based on data from two trials of PfSPZ vaccines in Africa where protection was markedly diminished in participants with parasitemia prior to clearance two weeks before immunization. We plan to extend the interval between pre-treatment and immunization from 2 to 5-6 weeks before the first immunization, to provide more time for the immune system to recover from the effects of parasitemia. Because immunization will be done during the dry season when malaria is rarely transmitted, only a few retreatments (if any) may be required, despite the 5- to 6-week gap, prior to the first vaccination. For the first immunization (V1), group 1 will receive one dose of vaccine (4x10^5PfSPZ) and groups 2 and 3 will receive one dose of normal saline (normal saline placebo). Four weeks later, group 1 will receive a second dose of vaccine (4x10^5 PfSPZ), group 2 will receive a first dose of vaccine (6x10^5 PfSPZ) and group 3 will receive a second dose of normal saline.

A syringe of vaccine and a syringe of normal saline are indistinguishable, facilitating the double-blind design. All administrations will be by DVI, a nearly painless procedure in which a narrow gauge needle is inserted into a superficial vein, blood flashback is demonstrated, and the contents of the syringe rapidly injected. Safety monitoring: Monitoring for adverse events (AEs) will take place during the 28-day interval between immunizations and for 28 days after the second immunization (56 days in total). Local (site of injection) AEs will be solicited for two days, systemic AEs will be solicited for 14 days and unsolicited AEs will be collected for 28 days after each immunization. In addition, participants will be instructed to notify the clinical team day or night should symptoms suggestive of malaria develop. Any symptoms consistent with malaria will be immediately investigated by TBS, which will be repeated if symptoms are ongoing - daily if the initial TBS is negative and symptoms are grade 1 or 2 in severity, or every 8 to 12 hours if initial TBS is negative and symptoms are grade 3 in severity. Malaria signs and symptoms include fever (axillary temperature in > 37.5°C [>99.5°F]), subjective fever, headache, dizziness, malaise, fatigue, chills, rigors, sweats, myalgia, arthralgia, nausea, vomiting, diarrhea, abdominal pain, cough and chest pain. Finally, medically-attended adverse events (MAAEs) and serious adverse events (SAEs) will be monitored throughout the trial. Laboratory tests (white blood count, neutrophil count, lymphocyte count, hemoglobin, platelets, creatinine, alanine aminotransferase) will be done on the day of each immunization and 7 days after each immunization.

Surveillance for malaria: Two weeks following immunization, active and passive surveillance for clinical malaria and malaria infection will begin. Passive detection will be achieved by encouraging all participants to immediately report any signs or symptoms consistent with malaria to the clinical team, which will be available 24/7. A TBS will be obtained as quickly as possible and read. A positive result will mark a clinical malaria endpoint, assuming that the case definition is met. It will also signify a malaria infection endpoint.

Active surveillance will consist of obtaining a TBS every two weeks from the entire study cohort starting two weeks after the second immunization, regardless of symptoms. These will be read in real-time only if there are malaria signs and symptoms. At each two week visit, participants will be reminded of the importance of contacting the clinical team if they develop malaria symptoms. The primary efficacy endpoint will be after 24 weeks of surveillance (26 weeks after immunization). Efficacy will also be calculated after the full 40 weeks of follow-up. A complete blood count will also be obtained at 24 weeks to see if vaccination with PfSPZ-LARC2 Vaccine had any effect on hemoglobin concentrations at the end of the rainy season.

TBS collected actively from asymptomatic individuals will be read retrospectively, and any new onset asymptomatic infections will be added as malaria infection endpoints as long as there was no clinical malaria endpoint reached in the same participant within two weeks of the asymptomatic parasitemia identified by active case detection.

Surveillance will continue past the 24 week primary endpoint until at least 40 weeks, with an option to continue for a second season of surveillance if merited by efficacy demonstrated during the first rainy season and identification of funding for additional follow-up. If there is no continuation, the last study visit will be at 40 weeks of surveillance (42 weeks after second immunization). At each two week visit when blood is sampled for TBS and at any time that TBS is made for the purpose of diagnosing clinical malaria, dried blood spots will be collected for possible later analysis by qPCR as an exploratory objective.

Prior to treating any malaria infection, blood samples will be obtained to allow for conducting genetic analyses of parasites, which could include sieve analysis to determine if lack of protection by vaccination is associated with particular genetic variants.

After treatment for malaria, 28 days of person-time at risk will be discounted (because of protection afforded by piperaquine), and then surveillance will continue to collect data on any additional parasitemias or clinical cases.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females, based on clinical and laboratory findings
2. From the age 18 to 50 years
3. Adults with a Body Mass Index (BMI) 18 to 30 Kg/m2.
4. Residence in the study area for the duration of the study.
5. Agreement to release medical information and to inform the study doctor concerning contraindications for participation in the study.
6. Willingness to be attended to by a study clinician and take all necessary medications prescribed during study period.
7. Agreement to provide contact information of a third party household member or close friend to study team.
8. Agreement not to participate in another clinical trial during the study period.
9. Agreement not to donate blood during the study period (until final clearance is completed)
10. Able and willing to complete the study visit schedule over the study follow up period.
11. Willingness to undergo HIV, hepatitis B (HBV), hepatitis C (HCV), and sickle cell anemia tests.
12. Volunteer participant can demonstrate their understanding of the study by responding correctly to 18 out of 20 true/false statements (in a maximum of two repeat attempts for those who failed to pass in the first attempt).
13. Signed written informed consent, in accordance with local practice.
14. Has not been treated with any antimalarial medication for at least two weeks prior to the initial clearance treatment.
15. Female volunteers aged 18 years and above must be non-pregnant (as demonstrated by a negative urine pregnancy test), and provide consent / assent of their willingness to take protocol-defined measures not to become pregnant during pre-treatment and immunization period and until 28 days after the second immunization. Acceptable measures to not become pregnant include oral or implanted contraceptives, IUD, abstinence, sterilization or sterile sexual partner. Women with a history of surgical or chemical sterilization (e.g., tubal ligation, hysterectomy, other) must provide written documentation of the procedure from a health care provider.
16. Demonstration of the ability to complete pre-vaccination drug clearance without significant untoward effects.

Exclusion Criteria:

1, Unable to provide informed consent including inability to pass the test of understanding.

2. Receipt of a malaria vaccine in a prior clinical trial. 3. History of a splenectomy or sickle cell disease. 4. History of a neurologic disorder (including non-febrile seizures or complex febrile seizures) or formal history of migraine headache.

5. Current use of systemic immunosuppressant pharmacotherapy. 6. Receipt of a live vaccine within 4 weeks of ﬁrst immunization or of 3 or more non-live vaccines within 2 weeks of ﬁrst immunization.

7. Women who are breast-feeding, pregnant or planning to become pregnant during the study period.

8. Known allergy to artemether-lumefantrine (AL), dihydroartemisinin-piperaquine (DHA-P), or any component of the investigational products.

9. History of anaphylaxis or other life-threatening reaction to a vaccine. 10. Participation in any study involving investigational vaccine or drug within 4 weeks prior to enrollment that in the estimation of the site PI might adversely aﬀect the individual's safety or the quality of data to be collected.

11. Evidence of increased cardiovascular disease risk; deﬁned as >10% ﬁve-year risk by non-laboratory method (Gaziano, 2008).

12. Plan to participate in another investigational vaccine/drug research during the study.

13. Plan for major surgery between enrollment until last study visit. 14. Use or planned use of any drug with anti-malarial activity that is not speciﬁed by the protocol.

15. Anticipated use of medications known to cause drug interactions with DHA-P (antiarrhythmics, neuroleptics, macrolide antibiotics, fluoroquinolones, imidazole and triazole antifungal agents, quinine, halofantrine, pentamidine and saquinavir, certain non-sedating antihistamines, all of which can aﬀect QT intervals ) or AL (the same list of drugs aﬀecting QT intervals plus rifampin, carbamazepine, phenytoin, St. John's wort and antiretroviral drugs).

16. Positive HIV, HBsAg or HCV serology. 17. History of or evidence for other chronic disease conditions including cancer, diabetes, renal failure, hypertension, tuberculosis, etc.

18. History of arrythmias or cardiac disease, or an abnormal electrocardiogram, deﬁned as one showing prolonged QT interval, pathologic Q waves and signiﬁcant ST-T wave changes; left ventricular hypertrophy; any non-sinus rhythm including isolated premature ventricular contractions, but excluding isolated premature atrial contractions; right or left bundle branch block; or advanced (secondary or tertiary) A-V heart block; or other clinically signiﬁcant abnormalities on the electrocardiogram. 19. Any clinically signiﬁcant deviation from the normal range in biochemistry or hematology tests measured at screening and not resolving (grade 1 abnormalities are allowed).

20. Any medical, psychiatric, social, behavioral or occupational condition or situation (including active alcohol or drug abuse aﬀecting social function) that, in the judgment of the site PI, impairs the participant's ability to give informed consent, increases the risk to the participant of participation in the study, aﬀects the ability of the participant to participate fully in the study, or might negatively impact the quality, consistency, integrity or interpretation of data derived from their participation in the study. 21. Inability to complete a course of malaria treatment prior to receipt of investigational product.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-04-04 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Vaccine efficacy of PfSPZ-LARC2 Vaccine as compared to normal saline, placebo against first Pf infection as detected by thick blood smear (TBS). | 2-24 weeks after last dose of vaccine or placebo
  TBS positive for asexual Pf at any parasite density collected every 2 weeks and at any time participants present with symptoms of malaria, starting 2 weeks after last dose of vaccine or placebo and extending 24 additional weeks.

SECONDARY OUTCOMES:
Safety and tolerability of PfSPZ-LARC2 Vaccine - solicited AEs | 14 days post each administration of vaccine or placebo
  Incidence of grade 3 solicited adverse events (AEs) in the 14 days post each administration of vaccine or placebo
Safety and tolerability of PfSPZ-LARC2 Vaccine- laboratory abnormalities | 1 week post each administration of vaccine or placebo
  Incidence of laboratory abnormalities at 1 week post each administration of vaccine or placebo
Safety and tolerability of PfSPZ-LARC2 Vaccine- unsolicited AEs | 28 days post each administration of vaccine or placebo
  Incidence of related grade 3 unsolicited AEs in the 28 days post each administration of vaccine or placebo
Safety and tolerability of PfSPZ-LARC2 Vaccine- SAEs | After the first administration of vaccine or placebo until the end of the study
  Incidence of related serious adverse events (SAEs) after the first administration of vaccine or placebo until the end of the study
Safety and tolerability of PfSPZ-LARC2 Vaccine- break-through vaccine strain blood stage infections | after the first administration of vaccine or placebo until the end of the study
  Incidence of any break-through vaccine strain blood stage infections
Vaccine efficacy against naturally transmitted first Pf clinical malaria | 2 weeks after last dose of vaccine or placebo and extending 24 additional weeks.
  Assess incidence of clinical malaria (primary case definition): Positive TBS at any parasite density plus
  1. measured axillary temperature ≥ 37.5 degrees Celsius or history of fever in the last 24 hours; or
  2. at least two of the following symptoms/ symptom groups: headache; chills and/or rigors; malaise and/or fatigue; dizziness and/or lightheadedness; myalgias and/or arthralgias; or (c) meeting criteria for severe malaria.
Antibody responses following vaccination and their association with vaccine efficacy | Two weeks to 24 weeks after the last immunization
  Anti-Plasmodium falciparum (Pf) circumsporozoite protein (CSP) antibody levels measured by ELISA before immunization, at least two weeks and 24 weeks after the last immunization and the association of these levels with vaccine efficacy against Pf infection and/or Pf clinical malaria.

CONTACTS AND LOCATIONS:
Overall Officials: Sodiomon B Sirima, MD PhD, Principal Investigator — Groupe de Recherche Action en Sante

IPD SHARING:
Plan to Share IPD: No